CLINICAL TRIAL: NCT01442142
Title: Self-Regulation Treatment for Pediatric Obesity
Brief Title: A Study to Determine the Effectiveness of a Self-regulation Program to Treat Pediatric Obesity
Acronym: ROC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHC FRD 06-32; AHC FRD 06-32 (Other Grant/Funding Number: University of Minnesota)
Record Dates: First submitted 2011-08-02; First posted 2011-09-28 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-09

CONDITIONS: Obesity
Keywords: obesity; pediatric; childhood; overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Appetitie Awareness (Experimental): Parents and kids assigned to this group with learn about appetite awareness and to appropriately respond to their "hunger meter."
  Interventions: Behavioral: CAAT: Appetite Awareness
- Cue Reactivity and Sensitivity Training (Experimental): Parents and kids in this group learn about how external cues can lead to overeating and how to better respond to these cues.
  Interventions: Behavioral: CRST: Volcravo
- Combined CAAT/CRST (Experimental): In this 14 week intervention combining Children's Appetite Awareness Training (CAAT) and Cue Reactivity and Sensitivity Training (CRST), parents and kids learn about both internal hunger cues and external cues that can cause one to overeat. Skills to learn the internal hunger cues and better responses to external cues are taught.
  Interventions: Behavioral: Combined CAAT and CRST program
- Control (No Intervention): Between baseline and the post-intervention data collection point, no intervention is given. Participants are given a take home binder of intervention materials at that second data collection point; they have the option of reviewing the material prior to the final follow-up data collection point.

INTERVENTIONS:
Behavioral: CAAT: Appetite Awareness — Participants in this Children's Appetite Awareness Training (CAAT) group learn to get in touch with the internal cues of hunger - aka the "hunger meter" - and practice skills to get back in touch with these internal cues of true hunger and fullness. Sessions occur once a week for 8 weeks.
  Arms: Appetitie Awareness
Behavioral: CRST: Volcravo — Participants in this Cue Reactivity and Sensitivity Training (CRST) group learn about how external cues can affect when and how much we eat (aka "volcravo - the craving volcano"). Over 8 weekly sessions, they practice skills to ride out the cravings external cues can cause.
  Arms: Cue Reactivity and Sensitivity Training
Behavioral: Combined CAAT and CRST program — Participants meet weekly for 14 weeks to learn about both Children's Appetite Awareness Training (CAAT) and Cue Reactivity and Sensitivity Training (CRST) - i.e. appetite awareness and external cues that affect food intake.
  Arms: Combined CAAT/CRST

SUMMARY:
The objective of this study is to pilot test, evaluate and compare the effects of Cue Reactivity and Sensitivity Training (CRST) and Children's Appetite Awareness Training (CAAT) in 48 children aged 8-12 years old. The central hypothesis is that CRST and CAAT will reduce eating in the absence of hunger in overweight children immediately following treatment and 6-months post treatment.

The primary aim of this proposed study is to evaluate the efficacy and compare the effectiveness of Cue Responsivity and Sensitivity Training (CRST) or Children's Appetite Awareness Training (CAAT) in decreasing eating in the absence of hunger (EAH) in overweight children. Following this first intervention, a second intervention to determine the efficacy of a combination program (combined CAAT & CRST) will be implemented.

The secondary aim of this study is to evaluate change in the following related measures for both children and adults who participated in CRST, CAAT, and the combination program: BMI for age, food intake, perceptions of control over eating, and self-efficacy in managing high-risk food situations.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) greater than the 85%-ile
* child consumes 10%+ of daily caloric need during Eating in the absence of hunger (EAH) assessment
* child between the age of 8-12 at the time of the first data collection visit

Exclusion Criteria:

* non-English speaking
* history of eating disorder
* food allergies
* unavailable on days of intervention meetings
* current participation in a weight loss or maintenance program
* presence of any medical condition affecting weight or growth
* presence of any physical, emotional, or behavioral disability that would prevent participant from taking part in the weekly study visits or the three data collection visits.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2008-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the amount of calories consumed during the Eating in the Absence of Hunger assessment at 3 months | Baseline and 3 months

SECONDARY OUTCOMES:
Change from baseline in BMI-for-age at 3 months. | Baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, PhD, Principal Investigator — University of Minnesota, now Univ of CA, San Diego; Lisa J Harnack, DrPH, Principal Investigator — University of Minnesota; Carol Peterson, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Boutelle KN, Zucker N, Peterson CB, Rydell S, Carlson J, Harnack LJ. An intervention based on Schachter's externality theory for overweight children: the regulation of cues pilot. J Pediatr Psychol. 2014 May;39(4):405-17. doi: 10.1093/jpepsy/jst142. Epub 2014 Jan 23. PMID 24459240